CLINICAL TRIAL: NCT00968279
Title: Coronary CT Angiography Using 320-Row Volume CT in Patients With Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Marc Dewey, Charité
Other Study IDs: EA1/134/08
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Atrial Fibrillation
Keywords: Patients with atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atrial Fibrillation

SUMMARY:
The primary objective of this study is to analyze the diagnostic accuracy of coronary CT angiography using 320 simultaneous detector results in patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Suspected coronary artery disease based on clinical findings or findings on other noninvasive imaging tests and planned coronary angiography within the next 14 days.
* Able to understand and willing to sign the Informed CF.

Exclusion Criteria:

* Creatinine of above 2.0 mg/dl
* Age below 50 years
* Women of child bearing potential (no hysterectomy, no menopause, or menopause since less than 12 months) must demonstrate a negative pregnancy test performed within 24 hours before CT.
* Inability to hold the breath for 10 seconds

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation scheduled to undergo coronary angiography due to suspected coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2009-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dewey, MD, PhD, Principal Investigator — Charité
Locations (1):
- Charité, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Zimmermann E, Dewey M. Whole-heart 320-row computed tomography: reduction of radiation dose via prior coronary calcium scanning. Rofo. 2011 Jan;183(1):54-9. doi: 10.1055/s-0029-1245629. Epub 2010 Aug 19. PMID 20725881
- [Background] Dewey M, Zimmermann E, Deissenrieder F, Laule M, Dubel HP, Schlattmann P, Knebel F, Rutsch W, Hamm B. Noninvasive coronary angiography by 320-row computed tomography with lower radiation exposure and maintained diagnostic accuracy: comparison of results with cardiac catheterization in a head-to-head pilot investigation. Circulation. 2009 Sep 8;120(10):867-75. doi: 10.1161/CIRCULATIONAHA.109.859280. Epub 2009 Aug 24. PMID 19704093
- [Background] Dewey M, Oncel D, Oncel G, Tastan A. Coronary CT angiography in patients with atrial fibrillation. Radiology. 2008 Aug;248(2):701; author reply 701-2. doi: 10.1148/radiol.2482080062. No abstract available. PMID 18641260